CLINICAL TRIAL: NCT05825807
Title: Complexity and Specificity of Antiepileptic Drug Treatment and Adherence to Therapy in Adolescence. Pilot Study on Drug Perception and Factors That May Affect it
Brief Title: Adherence to Pharmacological Antiepileptic Treatment in Adolescence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 09/19
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Epilepsy; Treatment Adherence
Keywords: Adolescence; Antiepileptic therapy; Treatment Adherence; Perception
MeSH Terms: conditions — Epilepsy; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epilepsy and its drug treatment affect fundamental aspects of an adolescent's lifestyle and can have major consequences on self-esteem and sense of identity. For many adolescents it is difficult to live with epilepsy and medication is difficult to accept; the side effects of medication, in particular even small changes in mental status and somatic appearance, are particularly feared and poorly tolerated. While it is true that drug-resistant epilepsies exist (about 30% of cases), it is also true that there exists a pseudo-resistance to drug treatment which is due to inadequate administration or poor adherence to treatment. It is estimated that 21 to 42% of patients on antiepileptic treatment don't adhere to the prescribed therapy. The literature emphasizes that non-adherence to treatment is a crucial problem for people with epilepsy, and that the adolescent population is particularly at risk. As with any chronic drug therapy, the therapeutic relationship plays an important role in the treatment of epilepsy. In adolescence, the communication that occurs within the therapeutic relationship takes on peculiar and specific aspects that go beyond the acquisition of anamnestic data and of what is usually reported explicitly in the interview. Communication must be centered on the adolescent's need for independence. Appropriate communication can make the adolescent feel more supported and can encourage him or her to gain self-awareness and control on decisions regarding his or her illness. For the physician, knowledge of the adolescent's point of view is indispensable in order to provide all the necessary information in an appropriate, understandable, and acceptable way, while at the same time acting as a mediator of communication.

The objective of this project is to describe and analyze adolescents' perception of antiepileptic treatment, their awareness of the disease and of the need for drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy
* Age between 12 and 18 years
* On treatment with antiepileptic drugs for at least one year
* Able to understand and complete the questionnaire

Exclusion Criteria:

* Subjects with moderate to severe intellectual disability

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with epilepsy treated with antiepileptic drugs for at least one year
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-11-12 (Estimated); Study Completion 2024-11-12 (Estimated)

PRIMARY OUTCOMES:
To describe adolescent's perception of need for antiepileptic treatment | At baseline
  Evaluated by the Antiepileptic drugs (AED) Necessity scale (6 items evaluating the perceived personal need for antiepileptic drugs). Each item provides 5 possible answers (1=strongly disagree, 2=disagree, 3=uncertain, 4=agree, 5=strongly agree)
To describe adolescent's concerns about potential adverse effects of antiepileptic drugs | At baseline
  Evaluated by the Antiepileptic drugs (AED)-Concerns scale (10 items evaluating concerns about potential adverse effects of antiepileptic drugs). Each item provides 5 possible answers (1=strongly disagree, 2=disagree, 3=uncertain, 4=agree, 5=strongly agree)

SECONDARY OUTCOMES:
To identify clinical factors influencing adolescent's perception of need for antiepileptic treatment | At baseline
  Clinical factors will be collected and association with AED-Necessity scale will be evaluated with multivariate analysis
To identify sociodemographic factors influencing adolescent's perception of need for antiepileptic treatment | At baseline
  Sociodemographic factors will be collected and association with AED-Necessity scale will be evaluated with multivariate analysis
To identify clinical factors influencing adolescent's concerns about potential adverse effects of antiepileptic drugs | At baseline
  Clinical factors will be collected and association with AED-Concerns scale will be evaluated with multivariate analysis
To identify sociodemographic factors influencing adolescent's concerns about potential adverse effects of antiepileptic drugs | At baseline
  Sociodemographic factors will be collected and association with AED-Concerns scale will be evaluated with multivariate analysis

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Zanus, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided